CLINICAL TRIAL: NCT00177567
Title: Treatment of Geriatric Bipolar Mood Disorders: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010614
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Manic Depression; Elderly; Late-Life
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium Carbonate; Valproic Acid; Risperidone; Olanzapine; Paroxetine; Bupropion; Lamotrigine; Venlafaxine Hydrochloride; Tranylcypromine; Mirtazapine

INTERVENTIONS:
Drug: lithium carbonate
Drug: Depakote-ER
Drug: risperidone
Drug: olanzapine
Drug: paroxetine
Drug: bupropion
Drug: lamotrigine
Drug: venlafaxine
Drug: tranylcypromine
Drug: mirtazapine

SUMMARY:
The purpose of this study is to collect pilot data on the feasibility of recruiting, eliciting informed consent, assessing, treating, and following patients aged 60 and older with bipolar mood disorders.

DETAILED DESCRIPTION:
Study specific aims are:

* to establish a recruitment, referral, and collaborative network for elderly bipolar patients, in collaboration with the NIMH funded STEP-BD
* to establish an outpatient treatment clinic at the Bellefield Towers site of the NIMH funded Intervention Research Center for Late Life Mood Disorders
* to implement standardized care pathways compatible with STEP-BD treatment algorithms for mood stabilizing pharmacotherapy.
* to document short- and long-term treatment response with respect to affective symptoms, sleep, general life functioning, cognition, treatment-emergent side effects
* to establish the clinical infrastructure necessary for randomized controlled clinical trials and for clinical research training in bipolar mood disorders of late-life.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Bipolar Disorder
* Folstein Mini-Mental Status Exam score of 18 or higher

Exclusion Criteria:

* Medical condition that precludes the use of both lithium and depakote
* If mood disturbance is deemed an organic mood disorder (i.e., iatrogenic, secondary to medication)
* If refuse to designate someone who the study staff can contact about bipolar symptoms, concerns about the subject's health, in an emergency, and/or inability to reach the subject.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-07; Study Completion 2004-01

PRIMARY OUTCOMES:
The percent of subjects remitting from their index affective episode, the time to remission, the percent of partially and non-remitting patients, the incidence of relapse during continuation treatment, and of recurrence during maintenance treatment

SECONDARY OUTCOMES:
Measures of affective symptoms, functional status, side effects, and cognition tracked over acute, continuation, and maintenance phases of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Reynolds III, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsubrgh Medical Center, Pittsburgh, Pennsylvania